CLINICAL TRIAL: NCT05617508
Title: N-DOSE AD: A Dose Optimization Trial of Nicotinamide Riboside in Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Haraldsplass Deaconess Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 428878
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease; Dementia
Keywords: NAD metabolism; Mitochondria; Nicotinamide Riboside
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded placebo-controlled study. 80 participants randomized in 1:1:2 ratio to either: 1. Placebo (n=20), 2. NR 1000mg for 3 months (n=20), 3. Dose escalation group: NR 1000mg 1st month, NR 2000mg 2nd month, NR 3000mg 3rd month (n=40).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both participants and all investigators are blinded during the trial and during data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo, no active ingredients. Administered in capsule form twice daily for the duration of the trial (12 weeks).
  Interventions: Other: Placebo
- Dietary Supplement: NR 1000 mg group (Experimental): Nicotinamide Riboside (NR) 1000mg total daily. Administered in capsule form in doses of 500mg twice daily for the duration of the trial (12 weeks).
  Interventions: Dietary Supplement: Nicotinamide Riboside supplementation 1000mg daily in total
- Dietary Supplement: NR dose escalation group (Experimental): Nicotinamide Riboside (NR) dose escalation group: 1000mg NR daily in doses of 500mg twice daily (week 1 - week 4), 2000mg NR daily in doses of 1000mg twice daily (week 5 - week 8), 3000mg NR daily in doses of 1500mg twice daily (week 9 - week 12).
  Interventions: Dietary Supplement: Nicotinamide Riboside dose escalation (up to 3000 mg daily in total)

INTERVENTIONS:
Other: Placebo — Placebo capsules administered twice daily for a total of 12 weeks.
  Arms: Placebo
Dietary Supplement: Nicotinamide Riboside supplementation 1000mg daily in total — Nicotinamide Riboside supplementation 1000mg daily in total
  Other Names: Niagen; NR
  Arms: Dietary Supplement: NR 1000 mg group
Dietary Supplement: Nicotinamide Riboside dose escalation (up to 3000 mg daily in total) — Nicotinamide Riboside supplementation up to 3000mg daily in total
  Other Names: Niagen; NR
  Arms: Dietary Supplement: NR dose escalation group

SUMMARY:
The goal of this double-blinded placebo-controlled randomized trial is to determine the optimal dose of nicotinamide riboside (NR), in individuals with Alzheimer's disease (AD).

The main questions the N-DOSE AD trial aims to answer are:

What dose of nicotinamide riboside (NR) is required to achieve maximal cerebral nicotinamide adenine dinucleotide (NAD) increase, measured by 31P-magnetic resonance spectroscopy (MRS) or cerebrospinal fluid (CSF) metabolomics)?

What dose of nicotinamide riboside (NR) is required to achieve maximal alteration in the cerebral metabolism patterns, measured by fluorodeoxyglucose-positron emission tomography (FDG-PET)?

What dose of nicotinamide riboside (NR) will have optimal effect in the absence of unacceptable toxicity?

Participants will be asked to do participate in:

Clinical examinations

Cognitive assessments

Lumbar puncture

Magnetic resonance imaging - positron emission tomography (MRI-PET) scannings

Biosampling

They'll be given placebo, 1000 mg NR or escalating doses of NR (1000 mg - 2000 mg - 3000 mg) over 12 weeks.

DETAILED DESCRIPTION:
N-DOSE AD is a double-blinded placebo-controlled randomized trial aiming to determine the optimal biological dose (OBD) of nicotinamide riboside (NR), in individuals with Alzheimer's disease (AD).

Individuals with AD (n = 80) will be recruited starting November 2022. Participants will be randomized 1:1:2 to either placebo group (n = 20) or NR 1000mg daily (n = 20) for 12 weeks or to a dose-escalation group where NR 1000mg daily will be administered week 1-4, NR 2000mg daily week 5-8 and NR 3000mg daily week 9-12 (n =40). Both the participants and the investigators will be blinded.

* Primary Objective:

  -- To compare the effect of orally administered nicotinamide riboside (NR), escalated to 1500 mg twice per day (3000 mg/day) in the dose escalation group (DE-group) - versus stable dosing of 500 mg twice per day (1000 mg/day) in the dose-stable group (DS-group) on cerebral NAD levels, at week 12.
* Secondary Objectives:

  * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in cerebral NAD levels from baseline to weeks 4, 8 and 12.
  * To compare the effectiveness of orally administered nicotinamide riboside (NR) 1500 mg twice per day versus 500 mg twice per day in augmenting the NAD-metabolome in the central nervous system (CNS) at week 12.
* Safety Objectives

  -- To determine the safety and tolerability of NR at a dose of 1000 mg, 2000 mg, and 3000 mg per day in AD.
* Exploratory Objectives:

  * Neuroimaging
  * To compare the effect of orally administered NR in the DE-group versus DS-group on the NR related metabolic pattern (NRRP) expression at week 12.
  * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in NRRP expression from baseline to weeks 4, 8 and 12.
  * To compare the effect of orally administered NR DE-group versus DS-group on the AD-related pattern (ADRP) expression at week 12.
  * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in ADRP expression from baseline to weeks 4, 8 and 12.
  * Metabolism & molecular markers
  * To compare the effect of orally administered NR in the DE-group versus DS-group on the NAD metabolome* in the blood, urine and central nervous system (CNS) at week 12.
  * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in the NAD metabolome* in blood and urine from baseline to weeks 4, 8 and 12.
  * To compare the effect of orally administered NR in the DE-group versus DS-group on serum and CSF inflammatory markers at week 12.
  * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in serum inflammatory markers from baseline to weeks 4, 8 and 12.
  * Clinical - cognitive & non motor symptom severity, quality of life
  * To compare the effect of orally administered NR in the DE-group versus DS-group on clinical severity of AD symptoms at week 12.
  * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and change in clinical severity of AD symptoms from baseline to weeks 4, 8 and 12.
  * To compare the effect of orally administered NR in the DE-group versus DS-group on ADL severity in AD at week 12.
  * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and change in ADL scores in AD from baseline to weeks 4, 8 and 12.
  * To compare the effect of orally administered NR in the DE-group versus DS-group on depressive symptoms in AD at week 12.
  * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and depressive symptoms in AD from baseline to weeks 4, 8 and 12.
  * To compare the effect of orally administered NR in the DE-group versus DS-group on neuropsychiatric symptoms in AD at week 12.
  * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and change in neuropsychiatric symptoms in AD from baseline to weeks 4, 8 and 12.
* Hypothesis-generating or resource-dependent endpoints (may be reported in follow-up or secondary publications).

  * To compare the effect of orally administered NR in the DE-group versus DS-group on gene expression at week 12.
  * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in gene expression from baseline to weeks 4, 8 and 12.
  * To compare the effect of orally administered NR in the DE-group versus DS-group on protein expression at week 12.
  * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in protein expression from baseline to weeks 4, 8 and 12.
  * To compare the effect of orally administered NR in the DE-group versus DS-group on serum and CSF inflammatory markers at week 12.
  * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in serum inflammatory markers from baseline to weeks 4, 8 and 12.
  * To compare the effect of orally administered NR in the DE-group versus DS-group on histone acetylation in AD at week 12.
  * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in histone acetylation in AD from baseline to weeks 4, 8 and 12.
  * To compare the effect of orally administered NR in the DE-group versus DS-group on H3K27 and H4K16 histone acetylation in AD at week 12.
  * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in on H3K27 and H4K16 histone acetylation in AD from baseline to weeks 4, 8 and 12.
  * To compare the effect of orally administered NR in the DE-group versus DS-group on the genomic distribution of H3K27 and H4K16 histone acetylation in AD at week 12.
  * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in the genomic distribution of H3K27 and H4K16 histone acetylation in AD from baseline to weeks 4, 8 and 12.
  * To compare the effect of orally administered NR in the DE-group versus DS-group on folate and one-carbon metabolism in AD at week 12.
  * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in folate and one-carbon metabolism in AD rom baseline to weeks 4, 8 and 12.
  * To compare the effect of orally administered NR in the DE-group versus DS-group on methyl donors in AD at week 12.
  * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in methyl-donors in AD from baseline to weeks 4, 8 and 12.
  * To compare the effect of orally administered NR in the DE-group versus DS-group on DNA methylation at week 12.
  * To assess the dose-response relationship between NR dose (1000 mg, 2000 mg, 3000 mg per day) and changes in methyl-donors in AD from baseline to weeks 4, 8 and 12.
  * To compare the effect of orally administered NR in the DE-group versus DS-group on synthesis of neurotransmitters in AD at week 12.
  * Determine whether NR-therapy affects the gut microbiome in a dose-responsive manner at week 12.
  * To compare the effect of orally administered NR in the DE-group versus DS-group on the gut metabolome at week 12.
* Procedures:

All participants will attend study visits at Baseline, week 4, week 8 and week 12. The study visits will consist of the following:

Assessment by physician and study nurse involved in the study including The Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog), the Clinical Dementia Rating (CDR), Montreal Cognitive Assessment Test (MoCA), Trail Making Test (TMT), The Lawton Instrumental Activities of Daily Living Scale (IADL), The Physical Self-Maintenance Scale (PSMS), Montgomery-Asberg Depression Rating Scale (MADRS), the The Neuropsychiatric Inventory Questionnaire (NPI-Q)

A 31P-magnetic resonance spectroscopy (MRS), 1H-magnetic resonance spectroscopy (MRS) and fluorodeoxyglucose-positron emission tomography (FDG-PET) scan.

Physical examination and measurement of vital signs. Routine blood tests. Urine sample collection. Faecal sample collection at Baseline and week 12. Cerebrospinal fluid (CSF) collection will be performed at Baseline and week 12.

ELIGIBILITY:
Inclusion Criteria:

* The following condition must apply to the prospective patient at screening prior to receiving study agent:

  * Diagnosis of probable Alzheimer Disease (AD) according to the core clinical criteria updated in the National Institute on Aging (NIA) and Alzheimer's Association guidelines.
  * Biomarker evidence consistent with AD neuropathologic change, defined by cerebrospinal fluid (CSF) markers.
  * Diagnosed with AD within two years from enrollment.
  * Clinical Dementia Rating (CDR) 0.5-1 (inclusive) at enrollment.
  * Age 50 to 85 years (inclusive) at the time of enrollment.
  * A study partner (i.e. a family member or a friend) able to provide study data and assist the participant in the study drug administration, i.e. contact ≥ 3 times weekly.
  * Capacity to provide written informed consent for study participation defined as Montreal Cognitive Assessment (MoCA) score ≥ 16 or Mini Mental State Evaluation (MMSE) score ≥ 20. MMSE or MoCA must have been performed within 6 months prior to baseline. If there is any doubt regarding the participants capacity to give informed consent we will ask for an independent evaluation by a consultant clinician who is not associated with the N-DOSE AD study.
  * Cholinesterase inhibitors and memantine can be used if stable for 8 weeks prior to baseline visit.
  * Able to undergo lumbar puncture.
  * Able to undergo magnetic resonance imaging (MRI)

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

* Diagnosis of dementia other than probable AD.
* Comorbidity that precludes study participation or data interpretation.
* Any psychiatric disorder that would interfere with compliance in the study.
* Any severe somatic illness that would interfere with compliance and participation in the study.
* Use of high dose vitamin B3 supplementation within 30 days of enrollment.
* Metabolic, neoplastic, or other physically or mentally debilitating disorder at baseline visit.
* Current treatment with Oral Anti-coagulation Therapies
* Implants that preclude MRI examinations, e.g. DBS, pacemaker

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Cerebral NAD levels measured by 31P-MRS | 12 weeks for primary analysis. 4, 8 and 12 weeks for secondary analysis.
  Change in cerebral NAD/ATP-α ratio measured by 31 Phosphorus magnetic resonance spectroscopy (31P-MRS) in the posterior brain (encompassing the occipital, parietooccipital and posterior parts of the temporal cortex).

SECONDARY OUTCOMES:
CSF NAD or other metabolite of the NAD metabolome, measured by LC-MS | 12 weeks
  Change in the cerebrospinal fluid (CSF) levels of NAD or other metabolites of the NAD metabolome*, measured by LC-MS.

OTHER OUTCOMES:
Frequency and severity of adverse events | 12 weeks
  The between-visit difference in incidence of treatment-associated mild/moderate/severe adverse events (AEs)
Change in gene and protein expression levels related to lysosomal and proteasomal function | 12 weeks
  The between-visit change in gene and protein expression levels related to lysosomal and proteasomal function in whole blood, measured by RNA sequencing (RNAseq) and proteomics (LC-MS), respectively.
Change in levels of one carbon metabolism metabolites | 12 weeks
  The between-visit change in one carbon metabolism/methylation pathway metabolites. Measured by HPLC-MS metabolomics in whole blood and CSF.
Between-change in depressive symptoms, measured by Montgomery-Asberg Depression Rating Scale (MADRS) | 12 weeks
  MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
Between-visit change in neuropsychiatric symptoms, measured by Change in Neuropsychiatric Inventory brief questionnaire form (NPI-Q) | 12 Weeks
  The NPI-Q measures the burden of 12 neuropsychiatric symptoms of dementia: delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor disturbance, nighttime behaviors, and appetite/eating. Symptom severity is rated on a 3-point scale with higher scores indicating worse symptoms. Minimum score would be 0 and maximum score would be 36.
Between-visit change in the Physical Self-Maintenance Scale (PSMS) | 12 weeks
  The PSMS includes 6 items, testing the following areas: toilet use, eating, dressing, physical appearance, deambulation and bath. The PSMS ranges from 1 to 30, with higher scores indicating WORSE functioning.
Between-visit change in the Lawton Instrumental Activities of Daily Living (IADL) Scale | 12 weeks
  The IADL scale consists of 8 items providing information about telephone use, preparing food, shopping, doing daily household chores, doing laundry, using transport, medication managing, and managing money. Scores range from 0 (dependent) to 8 (independent).
The between-visit change in executive functioning measured by the Trail Making Test (TMT) | 12 weeks
  The TMT is a timed test and the goal is to complete the test as accurately and as quickly as possible. Raw scores are reported in seconds to complete the test. For Part B, an average score is 75 seconds and a deficient score is greater than 273 seconds.
Between-visit change cognitive function measured by the Montreal Cognitive Assessment (MoCA) scale | 12 weeks
  MoCA scale (minimum score = 0, maximum score = 30) and a dichotomized cut-off score for normality of 26 or over. High scores indicate less cognitive impairment than low scores.
The between-visit chang in Clinical Dementia Rating scale sum of boxes (CDR-SB) | 12 weeks
  The CDR integrates assessments from 3 domains of cognition (memory, orientation, judgment/problem-solving) and 3 domains of function (community affairs, home/hobbies, personal care). Following caregiver interview and systematic participant examination, the rater assigns a score describing the participant's current performance level in each of these domains of life functioning. The "Sum of boxes" scoring methodology (CDR-SB) sums the score for each of the 6 domains and provides a value ranging from 0 to 18 with higher scores indicating greater impairment. Positive change from baseline indicates greater impairment.
Determining the between-visit change in the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog 13) | 12 weeks
  The ADAS-Cog 13 is a psychometric instrument that evaluates memory, attention, reasoning, language, concentration, planning, executive function, and praxis using an 13-point AD Assessment Scale. It has a minimum score of 0 and a maximum severity score of 85, and a higher score indicates more impairment. A reduction in between-visit scores indicates an improvement in cognitive functions.
Change in levels of monoamine neurotransmitters in CSF | 12 weeks
  The between-visit difference in levels of monoamine neurotransmitters in CSF.
Change in genomic distribution of DNA methylation | 12 weeks
  The between-visit difference in genomic distribution of DNA methylation, measured by the Illumina Infinium MethylationEPIC Kit.
Change in levels of DNA methylation | 12 weeks
  The between-visit difference in levels of DNA methylation, measured by the Illumina Infinium MethylationEPIC Kit.
Change in levels of histone acetylation | 12 weeks
  The between-visit difference in levels of histone panacetylation, and levels of site specific histone acetylation in whole blood, measured by immunoblotting and chromatin immunoprecipitation sequencing (ChIPseq).
Change in genomic distribution of histone acetylation | 12 weeks
  The between-visit difference in genomic distribution of histone acetylation in whole blood, measured by immunoblotting and chromatin immunoprecipitation sequencing (ChIPseq).
Change in gut microbiome composition | 12 weeks
  The between-visit difference in gut microbiome composition, assessed by metagenomics in fecal samples.
Change in faecal metabolomics | 12 weeks
  The between-visit difference in fecal metabolomics, including fatty acid profiling
Change in levels of inflammatory cytokines in serum and CSF | 12 weeks
  The between-visit difference in levels of inflammatory cytokines in serum and CSF, measured using the ELISA method.

CONTACTS AND LOCATIONS:
Overall Officials: Kristoffer Haugarvoll, MD, PhD, Principal Investigator — Haukeland University Hospital
Locations (2):
- Norway (2):
  - Haraldsplass Deaconess Hospital, Bergen, Vestland
  - Haukeland University Hospital, Bergen, Vestland

DOCUMENTS (2):
  • Study Protocol (2025-08-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT05617508/Prot_000.pdf
  • Statistical Analysis Plan (2025-11-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT05617508/SAP_001.pdf